CLINICAL TRIAL: NCT06435234
Title: Construction of a Risky Sexual Behaviour Intervention Programme for College Students Based on BCW Theory
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rong Zhang (Other)
Responsible Party: Sponsor-Investigator, Rong Zhang, Principal Investigator, Harbin Medical University
Organization: Harbin Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HMUDQ20231116201
Record Dates: First submitted 2024-05-24; First posted 2024-05-30 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Unsafe Sex
Keywords: Risky sexual behavior; BCW; college students; intervention program; unsafe sex
MeSH Terms: conditions — Unsafe Sex

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental)
  Interventions: Behavioral: risky sexual behavior intervention
- control group (No Intervention)

INTERVENTIONS:
Behavioral: risky sexual behavior intervention — Intervening in risky sexual behaviors among college students
  Arms: intervention group

SUMMARY:
Using the intervention functions of Behavior Change Wheel (BCW) and BCTs, we constructed an intervention program for college students' risky sexual behaviors by combining literature analysis, qualitative research, Delphi's expert correspondence, and pre-experiment (20 students in the test group and 20 students in the control group). Before the intervention (T0) and at the end of the intervention (12 weeks, T1), we measured students' psychosexual health, social support, and sexual self-efficacy using relevant scales to ensure the effectiveness of the intervention. By clarifying the influencing factors of college students' risky sexual behaviors, the proposed intervention program for college students' risky sexual behaviors can effectively reduce the incidence of college students' risky sexual behaviors, improve the level of college students' psychosexual health, increase the level of social support, improve the sense of sexual self-efficacy, improve the level of risk perception, enhance the ability of risky decision-making, reduce the risky behaviors, and reduce the occurrence of adverse outcomes, thus providing a reference and reference for the prevention and control of college students' risky sexual behaviors. This will provide reference for the prevention and control of risky sexual behaviors among college students.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥16 years;
2. full-time undergraduate college students;
3. engaged in risky sexual behaviors (including multiple sexual partners, unprotected sex, and casual sex, and one of them is considered to have engaged in risky sexual behaviors) during their college years;
4. able to clearly recall and describe the incident;
5. signed an informed consent form

Exclusion Criteria:

1. not wanting to be asked sex-related questions;
2. being screened at the beginning of the semester using the Mental Health Survey and diagnosed by a psychiatrist as having a mental illness (schizophrenia, major depressive disorder, bipolar disorder)

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-29 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Sexual mental health | pre-intervention（T0）; At the end of the intervention（12 weeks, T1）
  Questionnaire on Sexual Mental Health of College Students.A total of 31 entries were made, each of which was scored using a Likert 5 scale (1=completely disagree, 5=completely agree), with 25 items scored positively and 6 items scored negatively.
  Total scores ranged from 31-155, with higher scores indicating lower levels of psychosexual health
Social Support | pre-intervention（T0）; At the end of the intervention（12 weeks, T1）
  Social Support Rating Scale for College Students.There are 17 entries in total. Each entry was scored on a Likert 5-point scale (1=very non-compliant, 5=very compliant), with a total score range of 17-85, with higher scores indicating that 5-point Likert scale (1=very poorly met, 5=very well met), with a total score ranging from 17-85, with higher scores indicating that college students received more social support
Sexual self-efficacy | pre-intervention（T0）; At the end of the intervention（12 weeks, T1）
  Sexual Self-Efficacy Scale.There are a total of 34 entries. The first five dimensions were each scored on a 5-point Likert scale (1=strongly disagree, 5=strongly agree), and the last two dimensions were each scored on a scale of 0 (never) to -4 (more than 5 times), for a total score of 130, with higher scores indicating higher sexual self-efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- Daqing City, Heilongjiang Province, Daqing, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No
Non-disclosure of study data due to ethical requirements and protection of subjects' privacy